CLINICAL TRIAL: NCT06647303
Title: Better Conversations for Better Informed Consent: A Pilot Study to Automate Surgeon Training and Evaluate Patient-Reported Outcomes
Brief Title: Improving Surgical Communication for Patients in Wisconsin
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-1354; A539750 (Other: UW Madison); Protocol Version 4/17/2025 (Other: UW Madison)
Record Dates: First submitted 2024-10-16; First posted 2024-10-17 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Surgeons; Surgical Procedure, Unspecified
Keywords: decision making; communication
MeSH Terms: conditions — Communication | interventions — Focus Groups; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Surgical candidate (Experimental): Participants who are undergoing surgical consultation
  Interventions: Other: Surveys
- Stakeholder Focus Group (Experimental): Participants have previous experience with surgery
  Interventions: Other: Focus Group
- Surgeons (Experimental): Surgeons from the University of Wisconsin-Madison Department of Surgery with an outpatient surgical clinic who treat adult patients at UW Health
  Interventions: Behavioral: Training on communication framework

INTERVENTIONS:
Behavioral: Training on communication framework — Surgeons will receive training on the Better Conversations framework
  Arms: Surgeons
Other: Focus Group — Participants will attend a focus group to discuss the survey instruments used in this study which will help with future study design
  Arms: Stakeholder Focus Group
Other: Surveys — Participants will complete surveys regarding the surgeon's communication skills
  Arms: Surgical candidate

SUMMARY:
The purpose of this study is to evaluate a new training program to support communication between surgeons and their patients. The goal of the training program is to help patients get the information they need to make treatment decisions that are right for them.

Participants will complete surveys, attend a focus group, or receive training on Better Conversations, depending on the type of participant.

DETAILED DESCRIPTION:
Observational research shows that surgeons translate informed consent and shared decision-making standards into an overly complicated technical explanation of the patient's disease and treatment, and an overly simplified narrative that surgery will "fix" the patient's problem. They omit critical information about the goals and downsides of surgery and struggle to actualize the patient's role in medical decisions, while unintentionally concealing professional expertise. "Better Conversations" is a novel communication framework designed to address these problems. With this framework, surgeons provide context about clinical norms, clearly establish the goals of surgery, and comprehensively delineate the downsides of surgery as experienced by the patient to generate a deliberative space for patients to consider whether surgery is right for them. This paradigm-shifting framework meets the legal and ethical standards for informed consent, supports deliberation, and allows patients to anticipate and prepare for the experience of surgery.

The present study supports optimization of surgeon training and study procedures (Phase II) that is needed before large scale testing and dissemination (Phase III). Although this intervention is evidence based, collaborative efforts are needed to ultimately test and disseminate a major clinical shift. The long-term goal is for every surgeon to use Better Conversations with every patient, every time. The present study has two main objectives: 1) To make the education program scalable with automated assessment and feedback to surgeons using audio recordings from their clinical conversations, and 2) to evaluate patient and family reported outcome measures regarding surgeon communication.

ELIGIBILITY:
Inclusion Criteria:

Surgeons:

* Surgeons from University of Wisconsin - Madison Department of Surgery who have an outpatient surgical clinic and treat adult patients at UW Health

Surgical candidates:

* Age 18 or older
* Present to an enrolled surgeon's clinic with a surgical problem
* Decision making ability
* Speak English

Stakeholders:

* Must have previous experience with surgery (within 10 years)
* Speak English

Exclusion Criteria:

Surgeons:

* Solely treat minors (under age 18)

Surgical candidates:

* Lacking decision making capacity
* Unable to speak English

Stakeholders:

* Unable to speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 580 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Effect of automated training program | Up to 4 years
  Specialists will train 10 surgeons, audio recording 150 surgical consultations with surgical candidates. 100 audio recordings will be used as a training set to develop an automated assessment and feedback program. 50 recordings will be used to measure fidelity to the intervention with a summative assessment. 10 additional surgeons will be trained using the automated training and researchers will audio record 150 more surgical consultations with surgical candidates. Automated feedback will be provided for 100 of the consultations and researchers will measure fidelity to the automated intervention with a summative assessment of 50 consultations. The effect of the automated training program will be tested by comparing summative assessments of surgeon performance between the two differently-trained groups. Summative assessments to identify strengths and weaknesses of the automated training program will be used to revise the training iteratively for future study.
Compare effectiveness of specialist-delivered training versus automated training on participant-reported measures of surgeon communication | Up to 4 years
  Researchers will compare surgical candidate participant survey results between surgeons who received specialist-delivered training versus those who received automated training.

OTHER OUTCOMES:
To identify survey measures that have a strong baseline variance, the number of participants who evaluate communication skills of the surgeon in the top 10 percentile of scoring | Up to 4 years
  Data from the "Feeling Heard and Understood", "Preparation for Decision Making Scale", and the "Consumer Assessment of Healthcare Providers and Systems (CAHPS) Surgical Care Survey" instruments will be collected from patient participants, scored, and compared for their ceiling effects. Survey scores will be transformed from 1-100 with higher scores indicating better surgeon communication. The number of participants with scores in the top 10 percentile (90-100) will be reported for each survey, surveys with higher numbers of participants in the top 10th percentile have less baseline variance.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret (Gretchen) Schwarze, MD, MPP, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://patientpreferences.org/